CLINICAL TRIAL: NCT02383914
Title: Prospective Multicenter Trial on Diagnostics and Outcome of Ruptures of the Subscapularis After Arthroscopic Refixation
Brief Title: Clinical Study on Diagnostics and Outcome of Ruptures of the Subscapularis After Arthroscopic Refixation
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, PD Dr. med. Thomas Tischer, Prof. Dr. med. Thomas Tischer, University of Rostock
Other Study IDs: Subscap-042014
Record Dates: First submitted 2014-05-06; First posted 2015-03-10 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Subscapularis Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subscapularis rupture

SUMMARY:
The purpose of the trial is to optimize the diagnostics of subscapularis tendon tears and as the circumstances require to found a new classification.

The prime objective is a comparison of the conclusive of the clinic check-up, the sonographic and magnetic resonance tomography findings.

The secondary objective is to detect the correlation of the outcome with the age , the gender, the pathogenesis and attendant injuries.

ELIGIBILITY:
Inclusion Criteria:

* patients, who have turned 18
* suspected subscapularis tendon rupture

Exclusion Criteria:

* disability to understand the trial
* intraoperative intact supbscapularis tendon
* pre-surgical operation of the affected shoulder
* tumor
* infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of the patients, who got the operative therapy (refixaton of the subscapularis tendon) inclusive the post- treatment and satisfy the criteria .
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Shoulder function (Constant Score) | 52 weeks post- operative

SECONDARY OUTCOMES:
Strength | 12 and 52 weeks post-operative
  Strength will be measured by a special force sensor
Rerupture Rate | 12 and 52 weeks post-operative
  Sonographic investigation of rerupture rate

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Clinic of the University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany